CLINICAL TRIAL: NCT02981277
Title: Transcricoid Injection Versus Spray as You go Method for Local Anaesthesia During Flexible Bronchoscopy: A Randomised Controlled Trial
Brief Title: Transcricoid Injection vs. Spray as You go Method for Local Anaesthesia During Bronchoscopy
Acronym: CRISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr. Karan Madan, MD, DM Assistant Professor, Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Transcricoid RCT
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Disease
Keywords: Bronchoscopy; Lignocaine
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcricoid (Active Comparator): Lignocaine delivery using transcricoid injection
  Interventions: Drug: Transcricoid injection
- Spray as You go (Active Comparator): Lignocaine delivery using spray as you go method
  Interventions: Drug: Spray as you go

INTERVENTIONS:
Drug: Transcricoid injection — Lignocaine delivery using Transcricoid Injection
  Arms: Transcricoid
Drug: Spray as you go — Lignocaine delivery using Spray as you go method
  Arms: Spray as You go

SUMMARY:
Flexible bronchoscopy is one of the most widely performed procedures for diagnosis of various bronchopulmonary diseases. Most patients tolerate the procedure well although cough is often reported as a distressing symptom. It is likely that the acceptance of bronchoscopy would be significantly improved with control of cough. Use of sedation during bronchoscopy has been reported to improve procedure tolerance. However, awake(no sedation) bronchoscopy is routinely performed at many centres including ours.

Topical lignocaine is administered during bronchoscopy for local anaesthesia. There is limited literature on the efficacy of transtracheal/transcricoid injection versus spray as you go method for lignocaine delivery to the airways during bronchoscopy. This study would help to determine the procedure comfort for the patient while using the transtracheal/transcricoid method vs the spray as you go method.

DETAILED DESCRIPTION:
For all patients meeting the inclusion criteria, the demographic profile including age, sex, weight, smoking history and the type of procedures performed during bronchoscopy shall be recorded. A written informed consent will be obtained from all participants. The patients who undergo flexible bronchoscopy would be randomised in a one is to one ratio either to transcricoid or spray as you go group. Prior to the bronchoscopy blood pressure, pulse rate, respiratory rate and pulse oximetry saturation will be recorded at the baseline Patients in both the groups shall be prepared in a similar fashion except for the initial route of lignocaine delivery.

During the procedure, 1.5 ml aliquots of 2% lignocaine solution will be delivered through the bronchoscope when using spray-as-you go technique. Patients in the transcricoid group shall initially receive 5 ml of 2% lignocaine solution instilled transtracheally along with two baseline 1.5 cc bronchial spray aliquots of lignocaine, and additional aliquots of 2% lignocaine using the spray as you go method. The total lignocaine dose during the procedure will be recorded. The patients would be monitored for any adverse effects throughout the procedure. The bronchoscopist doing the procedure will be provided 2 VAS charts to mark the severity of cough and overall procedure satisfaction. Cough count shall be noted.

ELIGIBILITY:
Inclusion Criteria:

* Indication for diagnostic or therapeutic flexible bronchoscopy
* Age > 18 years
* Hemodynamic stability (defined as systolic BP >100 mm Hg and, <180 mm Hg).

Exclusion Criteria:

* Refusal of consent
* Known documented hypersensitivity to lignocaine
* Procedure performed under general anaesthesia
* Pregnancy
* Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3
* Bronchoscopy done through endotracheal or tracheostomy tube
* Midline neck mass or thyroid enlargement making the identification of cricothyroid membrane difficult'
* Patients with central airway obstruction
* Patients with active ongoing hemoptysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Cough count from bronchoscope introduction till reaching the carina | At study completion approximately 12 months

SECONDARY OUTCOMES:
Time from scope insertion to crossing the vocal cords | At study completion approximately 12 months
Overall procedure duration | At study completion approximately 12 months
Total Lignocaine dose | At study completion approximately 12 months
Operator rated overall procedure satisfaction | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, MD, DM, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided